CLINICAL TRIAL: NCT05735665
Title: Comparison Between Bowel Ultrasound-based Treat to Target Versus Routine Treat to Target Strategies in Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Mariangela Allocca, Gastroenterologist, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: T2T
Record Dates: First submitted 2023-01-27; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Ulcerative Colitis Chronic Moderate; Ulcerative Colitis Chronic Severe
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group: the bowel Ultrasound-based treat to target arm (Experimental): At W12 ± 4 and W24 ± 4, subjects will perform FC and bowel US and PRO will be recorded.
  If rectal bleeding > 2 + stool frequency > 2 AND FC > 250 mcg/g AND/OR MUC > 6.2, treatment will be changed according to GCP and international guidelines.
  Interventions: Diagnostic Test: bowel ultrasound
- control group: the routine Colonoscopy treat to target arm. (Other): At W12 ± 4 and W24 ± 4, subjects will perform FC and PRO will be recorded for all patients.
  If rectal bleeding > 2 + stool frequency > 2 AND FC > 250 mcg/g, treatment will be changed according to GCP and international guidelines. If rectal bleeding > 0 + stool frequency > 2 AND FC will be ≥ 50 mcg/g and ≤ 250 mcg/g, a RSS will be done in order to decide any treatment switch.
  Interventions: Diagnostic Test: colonoscopy

INTERVENTIONS:
Diagnostic Test: bowel ultrasound — Bowel US is a non-invasive tool which is able to measure intestinal inflammation by the use of emission of US from a specific probe. It is used externally, just moving the probe on the skin of the patient along the abdominal section. It does not require any contrast. The preparation used is just a fasting period of 6 hours.
  Arms: study group: the bowel Ultrasound-based treat to target arm
Diagnostic Test: colonoscopy — Colonoscopy is an endoscopic procedure where a tube is inserted from the anus up to the ileum of the patient. It requires bowel cleansing with polyethilenglicole up to 4 liters (depending on the preparation and the desired grade of cleansing) the day before the examination. Because it may be painful, usually sedation is provided.
  Arms: control group: the routine Colonoscopy treat to target arm.

SUMMARY:
UC (UC) is a chronic, relapsing and destructive inflammatory disorder of the colon which can lead to organ damage and impair quality of life.

Consensus guidelines recommend to go beyond resolution of clinical symptoms and achieve endoscopic remission. This long-term treatment goal in UC is commonly defined by a Mayo endoscopic subscore < 13, and is associated with prolonged clinical remission, lower rates of hospitalization and lower rates of colectomy. However, colonoscopy is an invasive and expensive procedure, unpleasant to patients, not without risks, especially during severe flares. Moreover, CS is time-consuming and expensive for the Healthcare System.

Clinical symptoms correlate well with endoscopic findings, and their improvement together to normalization of FC, are currently considered the short-term and intermediate-term targets to achieve. However, while asymptomatic patients with FC < 50 mcg/g have < 5% probability to have endoscopic lesions, and conversely patients with evident rectal bleeding and persistent increased stool frequency (> 3 stools above baseline) with FC > 250 mcg/g have less than 5% chance to have endoscopic remission, in patients in the intermediate scenarios with stool frequency score (SFS) 2 or 3 or rectal bleeding score (RBS) > 0, with FC values between 50 and 250 mcg/g, the uncertainty increases and CS should not be avoided.

Bowel US is a well-tolerated, non-invasive, patient friendly, cheap, easy-to-use tool to manage UC patients in clinical practice8. In addition, its ability to be performed as point-of-care bowel US may drastically change frequency of the assessment of treatment response, speeding the clinical decision-making process9. Recently, the investigators developed and externally validated non-invasive ultrasonography based criteria [Milan ultrasound criteria (MUC)] to assess and grade endoscopic activity in UC10,11. The investigators also confirmed that a MUC score > 6.2 is a valid cut-off to discriminate endoscopic activity, defined by a Mayo endoscopic subscore > 1 Bowel US is a well-tolerated, non-invasive, patient friendly, cheap, easy-to-use tool to manage UC patients in clinical practice. In addition, its ability to be performed as point-of-care bowel US may drastically change frequency of the assessment of treatment response, speeding the clinical decision-making process. Recently, the investigators developed and externally validated non-invasive ultrasonography based criteria [Milan ultrasound criteria (MUC)] to assess and grade endoscopic activity in UC14,15. The investigators also confirmed that a MUC score > 6.2 is a valid cut-off to discriminate endoscopic activity, defined by a Mayo endoscopic subscore > 1.

DETAILED DESCRIPTION:
Prospective interventional randomized open-label study to validate the role of US-based treat-to-target strategies in the decision-making process in patients with UC.

Patients seen at each participating center who are eligible for this study will be randomized 1:1 (computer generated randomization list) to enter one of two study arms up to Week 52:

1. study group: the bowel US-based treat to target arm
2. control group: the routine CS treat to target arm. At Week 52 ± 4, all patients in the two study arms will undergo CS, bowel US, PRO and FC as indicated for the screening phase.

Patients will be followed up and will undergo the study procedures as described below:

Bowel Ultrasound-based Treat to target arm At W12 ± 4 and W24 ± 4, subjects will perform FC and bowel US and PRO will be recorded.

If rectal bleeding > 2 + stool frequency > 2 AND FC > 250 mcg/g AND/OR MUC > 6.2, treatment will be changed according to the standard of care and international guidelines.

Routine CS Treat to target arm At W12 ± 4 and W24 ± 4, subjects will perform FC and PRO will be recorded for all patients.

If rectal bleeding > 2 + stool frequency > 2 AND FC > 250 mcg/g, treatment will be changed according to the standard of care and guidelines. If rectal bleeding > 0 + stool frequency > 2 AND FC will be ≥ 50 mcg/g and ≤ 250 mcg/g, a RSS will be done in order to decide any treatment switch.

The routine CS treat-to-target arm schedule is based on the recommendations of the STRIDE II. When appropriate, based on the investigator's judgement, CS can be replaced by a RSS.

Since the two strategies are part of the standards of care, no additional procedures outside the current clinical practice will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of UC since at least 8 weeks prior to inclusion
* Age ≥ 18 years
* Any gender/sex
* Active disease consistent with indication to start with systemic corticosteroids, biological agents or small molecules (defined as a patient-reported outcomes score, PRO > 2)
* Ability to understand and to comply with the study procedure and sign an informed consent form

Exclusion Criteria:

* Subjects with inflammation restricted to the rectum (≤ 15 cm from the anal verge);
* Subjects with severe UC (defined as a Mayo global score > 12, requiring hospitalization);
* Subjects with an endoscopic Mayo sub-score at baseline <2;
* Subjects with a MUC at baseline < 6.2;
* Pregnancy
* Subjects with any contraindication to any study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to evaluate the two strategies in terms of efficacy of bowel US-based strategy versus CS-based strategy in terms of remission. | 2 years
  Remission will be defined as global Mayo Score at week 52

CONTACTS AND LOCATIONS:
Overall Officials: MARIANGELA ALLOCCA, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Mariangela Allocca, Milan, Italy